CLINICAL TRIAL: NCT05249933
Title: The Efficiency of Pronase Granules in Gastric Cleaning of Magnetically Controlled Capsule Endoscopy: a Prospective Randomized Controlled Study
Brief Title: Pronase Granules in Gastric Cleaning
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Gastric preparation of MCE
Record Dates: First submitted 2022-02-09; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-02

CONDITIONS: Gastric Disease; Capsule Endoscopy
Keywords: capsule endoscopy; pronase granules; gastric preparation; visualization of gastric mucosa; randomized controlled study
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): All patients underwent a bowel preparation that consisted of a low-residue diet for 24 hours, fluid intake, and ingestion of two liters of polyethylene glycol-based electrolyte solution 12 hours before the examination. On the examination day, patients arrived at the hospital in the morning after an overnight fast (>8hours). Then they would be randomly assigned to the control group or pronase group randomly. 40 minutes before capsule ingestion, all patients swallowed 100ml clear water containing 50mg dimethicone. And 25 minutes before swallowing the capsule, the patient was asked to take 200ml warm water. There is still have 800-1000ml water for gastric filling 10 minutes before swallowing the capsule.
  Interventions: Drug: Deyou; Beijing Tide Pharmaceutical Co, China, containing 20,000 iu pronase granules combined with 1 g NaHCO3 to maintain the intragastric PH at 6-8
- Pronase group (Experimental): All patients underwent a bowel preparation that consisted of a low-residue diet for 24 hours, fluid intake, and ingestion of two liters of polyethylene glycol-based electrolyte solution 12 hours before the examination. On the examination day, patients arrived at the hospital in the morning after an overnight fast (>8hours). Then they would be randomly assigned to the control group or pronase group randomly. 40 minutes before capsule ingestion, all patients swallowed 100ml clear water containing 50mg dimethicone. And 25 minutes before swallowing the capsule, the patient was asked to take 20000 IU pronase Granules Combined with 1 g NaHCO3 dissolved in 200ml warm water to maintain the intragastric pH at 6 - 8. There is still have 800-1000ml water for gastric filling 10 minutes before swallowing the capsule.
  Interventions: Drug: Deyou; Beijing Tide Pharmaceutical Co, China, containing 20,000 iu pronase granules combined with 1 g NaHCO3 to maintain the intragastric PH at 6-8

INTERVENTIONS:
Drug: Deyou; Beijing Tide Pharmaceutical Co, China, containing 20,000 iu pronase granules combined with 1 g NaHCO3 to maintain the intragastric PH at 6-8 — Drink Deyo with 200ml warm water 25 minutes before swallowing the capsule to remove mucus in the stomach.

SUMMARY:
Magnetically controlled capsule endoscopy (MCE) is now widely used all over the world. However, the standard gastric preparation method by dimethicone we used clinically still has mucus at the bottom of the stomach. In this study, we aimed to determine whether pronase granules is helpful to improve the cleanliness of gastric mucosa in MCE.

DETAILED DESCRIPTION:
As a non-invasive and well-tolerated gastrointestinal examination method, magnetically controlled capsule endoscopy (MCE) is being increasingly used in different populations in recent years. Gastric preparation is extremely important for the completion rate (CR), image quality, and diagnostic efficiency because of the plica of gastric mucosa and the autonomous movement of the capsule in the gastrointestinal tract. After a series of explorations including air-producing powder, defoamer, protease preparation, patients are asked to drink about 800 ml-1000 ml water in a short time for standard gastric filling. However, the existing problems of gastric preparation such as abdominal distension, insufficient gastric filling, and long gastric retention time deserve attention. Different from the results of Zhu et al. (DLD, 2017), the current clinical experience shows that the addition of pronase granules in gastric preparation can often reduce the mucus in the stomach. But the standardized use of pronase granules remains to be further explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Those who underwent upper gastrointestinal and small intestinal mucosal examination under magnetically controlled capsule endoscopy at Shanghai Changhai Hospital and Chinese People's Liberation Army General Hospital after January 2020.
3. Able to provide informed consent.

Exclusion Criteria:

1. dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy, or post-abdominal radiation;
2. congestive heart failure, renal insufficiency, use of anticoagulant medication,
3. implanted metallic devices such as pacemakers, defibrillators, artificial heart valves or joint prostheses (although the low magnetic field used technically should not interfere with such devices);
4. pregnancy;
5. currently participating in another clinical study.
6. Patients who fail to follow the prescribed procedures for magnetically controlled capsule endoscopy;
7. Patients who only undergo gastric examination under magnetically controlled capsule endoscopy;
8. Patients who only undergo small bowel examination under magnetic control capsule endoscopy;
9. The patient's basic information in the database is incomplete#
10. Patient fail to be followed up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Gastric Cleanliness Score (GCS) | 2 weeks
  Six primary anatomical landmarks of the stomach (cardia, fundus, body, angulus, antrum, and pylorus) were recorded for evaluation. A 4-point grading scale was introduced to define the cleanliness as excellent (no adherent mucus and foam: score 4), good (mild mucus and foam but do not obscure vision: score 3), fair (considerable amount of mucus or foam present precluding a completely reliable examination: score 2) and poor (large amount of mucus or foam residue needing water to clear it: score 1). GCS was the total scores of all six landmarks, ranging from 6 (completely unprepared) to 24 (perfect). GCS of≥18 was regarded as acceptable.

SECONDARY OUTCOMES:
Visualization of the small bowel Visualization of the small bowel Visualization of the small bowel Visualization of the small bowel Visualization of the small bowel | 2 weeks
  Visualization of the small bowel was determined by the percentage of time during which the small-bowel view was clear, defined as not obscured more than 50% of the screen view. The clear-viewing percentage of the total small bowel transit time assessed by a 4-point scale :0, less than 25%; 1, 25% to 49%; 2, 50% to 75%; and 3, greater than 75%.
Fullness score | 2 weeks
  Fullness is the subjective feeling of patients assessed with visual analogue scale (VAS). VAS typically take the form of a straight line with two extreme states anchored at either end. In this study, it is a 100mm VAS with a question"How full do you feel?"anchored with "not at all full"at the left side and "as full as I have ever felt" at the right side. Patients will be asked to mark their feelings on the line. The distance (mm) between the far left and the marked point is the score of fullness. 0 represents no perception at all, 10 indicates pain and needs to be stopped immediately.
Gastric Examination Time (GET) | 2 weeks
  The time taken for the gastric examination to the endoscopist's satisfaction.
Esophageal transit time (ETT) | 2 weeks
  The time between the first image of esophagus and the first image of stomach.
Gastric transit time (GTT) | 2 weeks
  The time between the first image of stomach and the last image of stomach.
Small bowel transit time (SBTT) | 2 weeks
  The time between the last image of stomach and the image of ileocecal valve.
Completion Rate (CR) | 2 weeks
  The completion of stomach was defined as the observation of cardia, fundus, body, angulus, antrum and pylorus and the completion of small bowel examination was defined as the ileocecal valve was photographed.The completion rate in each group was defined as the percentage of patients with a complete examination out of the total number of patients examined.
Adverse events occurence rate | 2 weeks
  The safety were evaluated at two week after procedure for any adverse events such as infection, pain, nausea, vomiting and capsule impaction or retention.
Detection rate of lesions | 2 weeks
  The detection rate of lesions in different digestive part (esophagus, stomach, duodenum, small intestine) found by MCE.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu SG, Qian YY, Tang XY, Zhu QQ, Zhou W, Du H, An W, Su XJ, Zhao AJ, Ching HL, McAlindon ME, Li ZS, Liao Z. Gastric preparation for magnetically controlled capsule endoscopy: A prospective, randomized single-blinded controlled trial. Dig Liver Dis. 2018 Jan;50(1):42-47. doi: 10.1016/j.dld.2017.09.129. Epub 2017 Oct 6. PMID 29110963
- [Result] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Result] Krijbolder MS, Grooteman KV, Bogers SK, de Jong DJ. Addition of simethicone improves small bowel capsule endoscopy visualisation quality. Neth J Med. 2018 Jan;76(1):27-31. PMID 29380729
- [Result] Cave DR, Hakimian S, Patel K. Current Controversies Concerning Capsule Endoscopy. Dig Dis Sci. 2019 Nov;64(11):3040-3047. doi: 10.1007/s10620-019-05791-4. PMID 31468267
- [Result] Shamsudhin N, Zverev VI, Keller H, Pane S, Egolf PW, Nelson BJ, Tishin AM. Magnetically guided capsule endoscopy. Med Phys. 2017 Aug;44(8):e91-e111. doi: 10.1002/mp.12299. Epub 2017 Jun 23. PMID 28437000
- [Result] Jiang X, Pan J, Li ZS, Liao Z. Standardized examination procedure of magnetically controlled capsule endoscopy. VideoGIE. 2019 May 30;4(6):239-243. doi: 10.1016/j.vgie.2019.03.003. eCollection 2019 Jun. No abstract available. PMID 31194028